CLINICAL TRIAL: NCT07023653
Title: Comparison of Clinical Outcomes Between All-Inside and Complete Tibial Tunnel Techniques in Anterior Cruciate Ligament Reconstruction Among Patients With ACL Ruptures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Andri Maruli Tua Lubis, Prof. Dr. Andri M.T. Lubis, MD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-07-0995
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: All-inside Techniques
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- All-Inside Technique (Active Comparator): Patients With ACL Ruptures will undergo ACL reconstruction surgery with All-inside techniques
  Interventions: Procedure: All-Inside Techniques
- Complete Tibial Tunnel (Active Comparator): Patients With ACL Ruptures will undergo ACL reconstruction surgery with complete tibial tunnel techniques
  Interventions: Procedure: Complete Tibial Tunnel techniques

INTERVENTIONS:
Procedure: All-Inside Techniques — All-inside ACL reconstruction technique avoids creating full-length bone tunnels. Instead, it uses retrograde drilling to form bone sockets, and the graft is secured with adjustable-loop suspensory fixation on both the femur and tibia.
  Arms: All-Inside Technique
Procedure: Complete Tibial Tunnel techniques — Complete Tibial Tunnel Technique is a conventional technique for ACL reconstruction which involves the creation of full-length bone tunnels in the tibia for graft passage via an anterograde approach. Graft fixation is typically achieved using a bio-interference screw on the tibial side and a fixed-loop suspensory device on the femoral side
  Arms: Complete Tibial Tunnel

SUMMARY:
This study aims to compare the functional outcomes of patients with ACL rupture following ACL reconstruction surgery using hamstring grafts, between the all-inside technique and the complete tibial tunnel technique. The hamstring graft, which serves as the tissue substitute for the damaged ACL, is harvested from the posterior thigh of the patient and used to replace the torn ligament during reconstruction

DETAILED DESCRIPTION:
This Study was conducted usingdouble blind randomized controlled trial (RCT), patients who agree to participate in the study will be randomized to undergo ACL reconstruction using either the All-inside technique or the complete tibial tunnel technique. Clinical outcomes, including tibial translation, pain severity, IKDC score, and Tegner score, will be evaluated through anamnesis and physical examination at the outpatient orthopedic clinic at 3, 6, 9, and 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with anterior cruciate ligament rupture
* Patients within the age range of 18 to 65 years

Exclusion Criteria:

* Patients with Multiple Ligament Injuries in the Knee Joint
* Patients with a pregnancy condition
* Patients with Severe Osteochondral Defect (ICRS 4)
* Patients with signs of inflamation in knee joint

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Tibial Translation | Before surgery, 3rd month, 6th month, 9th month, and 12 month after surgery
  Objective measurement of the anterior tibial translation relative to the femur will be performed using a rolimeter during the Lachman test.
Pain scale using Visual Analogue Scales | Before surgery, 3rd month, 6th month, 9th month, and 12 month after surgery
  Pain scale on the injured knee, where the minimum value is 0 = no pain, and the maximum value is 100 = severe pain. A higher scale means worse outcomes.
International Knee Documentation Comittee (IKDC) Score | Before surgery, 3rd month, 6th month, 9th month, and 12 month after surgery
  Knee Function Assessment
Tegner-Lysholm Score Knee Scoring Scale | Before surgery, 3rd month, 6th month, 9th month, and 12 month after surgery
  a tool to assess knee function
Hamstring Graft Diameter | Intra-operative
  The thickness of the hamstring graft after harvesting and folding will be measured using a sizing block with various intra-operative hole sizes

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. dr. Andri M.T. Lubis SpOT (K), Principal Investigator — Indonesia University
Locations (2):
- Indonesia (2):
  - Indonesian University Hospital, Depok
  - Cipto Mangunkusumo Hospital, Jakarta Pusat

REFERENCES:
- [Background] Kouloumentas P, Kavroudakis E, Charalampidis E, Kavroudakis D, Triantafyllopoulos GK. Superior knee flexor strength at 2 years with all-inside short-graft anterior cruciate ligament reconstruction vs a conventional hamstring technique. Knee Surg Sports Traumatol Arthrosc. 2019 Nov;27(11):3592-3598. doi: 10.1007/s00167-019-05456-9. Epub 2019 Mar 19. PMID 30888448
- [Background] Rahardja R, Zhu M, Love H, Clatworthy MG, Monk AP, Young SW. Effect of Graft Choice on Revision and Contralateral Anterior Cruciate Ligament Reconstruction: Results From the New Zealand ACL Registry. Am J Sports Med. 2020 Jan;48(1):63-69. doi: 10.1177/0363546519885148. Epub 2019 Nov 15. PMID 31730379
- [Background] Samitier G, Vinagre G. Hamstring Braid Graft Technique for Anterior Cruciate Ligament Reconstruction. Arthrosc Tech. 2019 Jul 19;8(8):e815-e820. doi: 10.1016/j.eats.2019.03.022. eCollection 2019 Aug. PMID 31696044
- [Background] Kennedy JC, Weinberg HW, Wilson AS. The anatomy and function of the anterior cruciate ligament. As determined by clinical and morphological studies. J Bone Joint Surg Am. 1974 Mar;56(2):223-35. No abstract available. PMID 4452683
- [Background] Girgis FG, Marshall JL, Monajem A. The cruciate ligaments of the knee joint. Anatomical, functional and experimental analysis. Clin Orthop Relat Res. 1975 Jan-Feb;(106):216-31. doi: 10.1097/00003086-197501000-00033. PMID 1126079
- [Background] Tan JL, Chang PC, Mitra AK, Tay BK. Anthropometry of anterior cruciate ligament in Singaporean Chinese. Ann Acad Med Singap. 1998 Nov;27(6):776-9. PMID 10101548
- [Background] Pontoh LA, Rahyussalim AJ, Widodo W, Fiolin J, Rhatomy S. Anthropometric study as a predictor of anterior cruciate ligament sizes in Asian Indonesian population. J Orthop Surg (Hong Kong). 2021 Jan-Apr;29(1):23094990211000462. doi: 10.1177/23094990211000462. PMID 33745362
- [Background] Brown JA, Brophy RH, Franco J, Marquand A, Solomon TC, Watanabe D, Mandelbaum BR. Avoiding allograft length mismatch during anterior cruciate ligament reconstruction: patient height as an indicator of appropriate graft length. Am J Sports Med. 2007 Jun;35(6):986-9. doi: 10.1177/0363546506298584. Epub 2007 Mar 2. PMID 17337725
- [Background] Denti M, Bigoni M, Randelli P, Monteleone M, Cevenini A, Ghezzi A, Schiavone Panni A, Trevisan C. Graft-tunnel mismatch in endoscopic anterior cruciate ligament reconstruction. Intraoperative and cadaver measurement of the intra-articular graft length and the length of the patellar tendon. Knee Surg Sports Traumatol Arthrosc. 1998;6(3):165-8. doi: 10.1007/s001670050093. PMID 9704323
- [Background] Meijer K, Saper M, Joyner P, Liu W, Andrews JR, Roth C. Minimizing Graft-Tunnel Mismatch in Allograft Anterior Cruciate Ligament Reconstruction Using Blumensaat's Line: A Cadaveric Study. Arthroscopy. 2018 Aug;34(8):2438-2443.e1. doi: 10.1016/j.arthro.2018.03.006. Epub 2018 May 3. PMID 29730211
- [Background] Chiang ER, Ma HL, Wang ST, Hung SC, Liu CL, Chen TH. Hamstring graft sizes differ between Chinese and Caucasians. Knee Surg Sports Traumatol Arthrosc. 2012 May;20(5):916-21. doi: 10.1007/s00167-011-1653-3. Epub 2011 Aug 25. PMID 21866349
- [Background] Tang SP, Wan KH, Lee RH, Wong KK, Wong KK. Influence of hamstring autograft diameter on graft failure rate in Chinese population after anterior cruciate ligament reconstruction. Asia Pac J Sports Med Arthrosc Rehabil Technol. 2020 Aug 12;22:45-48. doi: 10.1016/j.asmart.2020.07.005. eCollection 2020 Oct. PMID 32913712
- [Background] Colombet P, Graveleau N. An Anterior Cruciate Ligament Reconstruction Technique With 4-Strand Semitendinosus Grafts, Using Outside-In Tibial Tunnel Drilling and Suspensory Fixation Devices. Arthrosc Tech. 2015 Sep 28;4(5):e507-11. doi: 10.1016/j.eats.2015.05.014. eCollection 2015 Oct. PMID 26697313
- [Background] Takahashi T, Watanabe S, Ito T. A Surgical Technique for Anterior Cruciate Ligament Reconstruction Using Semitendinosus Graft: An All-Inside Transfemoral Approach. Arthrosc Tech. 2023 May 29;12(6):e975-e982. doi: 10.1016/j.eats.2023.02.035. eCollection 2023 Jun. PMID 37424637
- [Background] Jones PE, Schuett DJ. All-Inside Anterior Cruciate Ligament Reconstruction as a Salvage for Small or Attenuated Hamstring Grafts. Arthrosc Tech. 2018 Apr 9;7(5):e453-e457. doi: 10.1016/j.eats.2017.11.007. eCollection 2018 May. PMID 29868418
- [Background] Fritsch B, Figueroa F, Semay B. Graft Preparation Technique to Optimize Hamstring Graft Diameter for Anterior Cruciate Ligament Reconstruction. Arthrosc Tech. 2017 Nov 13;6(6):e2169-e2175. doi: 10.1016/j.eats.2017.08.011. eCollection 2017 Dec. PMID 29349014
- [Background] Rante SDT, Santoso A, Sibarani T, Utomo DN. All-inside vs. conventional method in anterior cruciate ligament (ACL) reconstruction: systematic review and meta-analysis. Indones J Biomed Sci. 2022;16(2):47-59.
- [Background] Lubowitz JH, Schwartzberg R, Smith P. Randomized controlled trial comparing all-inside anterior cruciate ligament reconstruction technique with anterior cruciate ligament reconstruction with a full tibial tunnel. Arthroscopy. 2013 Jul;29(7):1195-200. doi: 10.1016/j.arthro.2013.04.009. PMID 23809454
- [Background] Ashraf Y, Senevirathna SR, Ashraf T. Conventional versus 'all-inside' anterior cruciate ligament reconstruction: a randomized controlled trial comparing hamstring strength and functional outcome. Bone Jt Open. 2020 Nov 4;1(11):706-708. doi: 10.1302/2633-1462.111.BJO-2020-0012.R1. PMID 33241220
- [Background] Lubowitz JH, Ahmad CS, Anderson K. All-inside anterior cruciate ligament graft-link technique: second-generation, no-incision anterior cruciate ligament reconstruction. Arthroscopy. 2011 May;27(5):717-27. doi: 10.1016/j.arthro.2011.02.008. PMID 21663726
- [Background] Lubowitz JH. No-tunnel anterior cruciate ligament reconstruction: the transtibial all-inside technique. Arthroscopy. 2006 Aug;22(8):900.e1-11. doi: 10.1016/j.arthro.2006.06.003. PMID 16904591
- [Background] Morgan CD, Kalmam VR, Grawl DM. Isometry testing for anterior cruciate ligament reconstruction revisited. Arthroscopy. 1995 Dec;11(6):647-59. doi: 10.1016/0749-8063(95)90104-3. PMID 8679023
- [Background] Lin R, Zhong Q, Wu X, Cui L, Huang R, Deng Q, Zuo J, Jiang C, Li W. Randomized controlled trial of all-inside and standard single-bundle anterior cruciate ligament reconstruction with functional, MRI-based graft maturity and patient-reported outcome measures. BMC Musculoskelet Disord. 2022 Mar 26;23(1):289. doi: 10.1186/s12891-022-05231-x. PMID 35337306
- [Background] Ardern CL, Taylor NF, Feller JA, Webster KE. Return-to-sport outcomes at 2 to 7 years after anterior cruciate ligament reconstruction surgery. Am J Sports Med. 2012 Jan;40(1):41-8. doi: 10.1177/0363546511422999. Epub 2011 Sep 23. PMID 21946441
- [Background] Teng Y, Zhang X, Da L, Hu J, Wang H, Han H, Wu M, Zhang S, Xia Y. Whether sutures reduce the graft laceration caused by interference screw in anterior cruciate ligament reconstruction? A biomechanical study in vitro. BMC Musculoskelet Disord. 2021 Jun 22;22(1):571. doi: 10.1186/s12891-021-04457-5. PMID 34158018
- [Background] Goyal T, Das L, Paul S, Choudhury AK, Sethy SS. Outcomes of retro-drilled all-inside tibial tunnel vs complete tibial tunnel techniques in anterior cruciate ligament reconstruction-a comparative study. Eur J Orthop Surg Traumatol. 2022 Apr;32(3):523-532. doi: 10.1007/s00590-021-03011-2. Epub 2021 May 24. PMID 34028623
- [Background] Connaughton AJ, Geeslin AG, Uggen CW. All-inside ACL reconstruction: How does it compare to standard ACL reconstruction techniques? J Orthop. 2017 Mar 19;14(2):241-246. doi: 10.1016/j.jor.2017.03.002. eCollection 2017 Jun. PMID 28360487
- [Background] Bosco F, Giustra F, Ghirri A, Cacciola G, Masse A, Capella M. All-Inside Anterior Cruciate Ligament Reconstruction Technique: Tips and Tricks. J Clin Med. 2023 Sep 6;12(18):5793. doi: 10.3390/jcm12185793. PMID 37762734
- [Background] Evans S, Shaginaw J, Bartolozzi A. Acl reconstruction - it's all about timing. Int J Sports Phys Ther. 2014 Apr;9(2):268-73. PMID 24790787
- [Background] Samitier G, Marcano AI, Alentorn-Geli E, Cugat R, Farmer KW, Moser MW. Failure of Anterior Cruciate Ligament Reconstruction. Arch Bone Jt Surg. 2015 Oct;3(4):220-40. PMID 26550585
- [Background] Deviandri R, van der Veen HC, Lubis AMT, Postma MJ, van den Akker-Scheek I. Translation, Cross-Cultural Adaptation, Validity, and Reliability of the Indonesian Version of the IKDC Subjective Knee Form. Orthop J Sports Med. 2021 Sep 29;9(9):23259671211038372. doi: 10.1177/23259671211038372. eCollection 2021 Sep. PMID 34604432
- [Background] Deviandri R, van der Veen HC, Lubis AMT, Utoyo GA, van den Akker-Scheek I, Postma MJ. Burden and Cost of Anterior Cruciate Ligament Reconstruction and Reimbursement of Its Treatment in a Developing Country: An Observational Study in Indonesia. Clinicoecon Outcomes Res. 2022 Jul 17;14:479-486. doi: 10.2147/CEOR.S368840. eCollection 2022. PMID 35872972